CLINICAL TRIAL: NCT00209352
Title: Randomized Trial of Long-Term Oral Acyclovir Usage to Prevent Varicella Zoster Virus Infection After Allogeneic Bone Marrow Transplant
Brief Title: Long-Term Oral Acyclovir Usage to Prevent Herpes Zoster Virus Infection After Bone Marrow Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Burroughs Wellcome (Industry); National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: FHCRC IR 420; CA 18029; CA 15704; Burroughs Wellcome Fund; FHCRC Protocol 236.00
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: VZV Infection After Bone Marrow Transplantation
Keywords: Varicella Zoster Virus Infection; VZV infection; Oral Acyclovir; Allogeneic Bone Marrow Transplantation; Allogeneic Hematopoietic Cell Transplantation
MeSH Terms: conditions — Varicella Zoster Virus Infection | interventions — Acyclovir

INTERVENTIONS:
Drug: Acyclovir

SUMMARY:
The objective of this study is to prevent reactivation of herpes zoster during the first year after transplant.

DETAILED DESCRIPTION:
Herpes zoster infection occurs in 30% of allogeneic hematopoietic cell transplant (HCT) recipients who had a history of varicella zoster virus (VZV) infection. A safe and effective prevention strategy has not been established.

77 marrow allograft recipients at risk for VZV reactivation were randomized to oral acyclovir 800 mg twice daily or placebo given from day 30 until day 365 and were followed for toxicity and clinical evidence of herpes zoster infection.

ELIGIBILITY:
Inclusion Criteria:

* 10 years or older
* Both sex (male or female)
* Allogeneic transplant patient for hematologic malignancy or aplastic anemia

Exclusion Criteria:

* Previous intolerance to acyclovir
* Patients who are unavailable for follow-up
* Patients in whom drug compliance may be a problem
* Evidence of active VZV infection
* VZV infection in the initial 1 month after transplant
* Pregnant women, lactating women, or those not using adequate contraception
* Creatinine > 3.0 mg/dl.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1985-06; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
VZV infection at one year

SECONDARY OUTCOMES:
VZV infection after discontinuation of prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boeckh, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Result] Boeckh M, Kim HW, Flowers ME, Meyers JD, Bowden RA. Long-term acyclovir for prevention of varicella zoster virus disease after allogeneic hematopoietic cell transplantation--a randomized double-blind placebo-controlled study. Blood. 2006 Mar 1;107(5):1800-5. doi: 10.1182/blood-2005-09-3624. Epub 2005 Nov 10. PMID 16282339